CLINICAL TRIAL: NCT03483831
Title: Effects of Hydration Status on Cognitive Performance in Adolescents Aged 12-14
Brief Title: Hydration Status and Cognitive Performance in Adolescents
Acronym: SMARTH2O
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Policlinico S. Donato (Other)
Responsible Party: Principal Investigator, Alexis Elias Malavazos, Leader of the High Speciality Center for Dietetics, Nutritional Education and Cardiometabolic Prevention, IRCCS Policlinico S. Donato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FLUIDA-MENTE
Record Dates: First submitted 2018-03-12; First posted 2018-03-30 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Hydration Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Students of 5 secondary school classes aged 12-14
  Interventions: Behavioral: Intervention group
- Control group (No Intervention): Students of 5 secondary school classes aged 12-14

INTERVENTIONS:
Behavioral: Intervention group — Refillable water dispensers will be placed in each class of the intervention group to facilitate water access: every class will receive 5 bottles (18 Liters/each) per week for a total of 5 months. Every student will receive a re-usable water bottle.
  Arms: Intervention group

SUMMARY:
Objective: to evaluate hydration status and his impact on cognitive performance in adolescents-based cohort study.

Methods: A randomized controlled pilot study is active in ten classes of one middle school (n=214 adolescents aged 12-14; including dismissed students) in an urban area around Milan, five classes being assigned to the intervention group and five classes to the control group. The five school-months intervention (from January to May 2018) includes changes in class environment (water dispenser to refill constantly, re-usable water bottles and educational posters about water consumption) and individual reinforcement tools (text messages and school lessons). The main endpoint is going to be the hydration status with osmolality urine test (dehydration status≥800 mOsm/kg). The secondary endpoint is going to be the correlation between the hydration status and cognitive performance (attention, short-term memory and concentration) through administration of neuropsychological tests from Neuropsychological Assessment Battery for Adolescence (BVN 12-18).

Results: it is expected an improvement of hydration status in intervention group versus control group and positive effects of a correct hydration on cognitive performance.

DETAILED DESCRIPTION:
INTRODUCTION Energy metabolism is higher per kilogram body weight in children than in adults. 1 Children aged from 11 to 14 should consume at least 1.5 liters of water per day, according to EFSA advice (European Food Safety Authority) 2.

This amount of daily water is difficult to reach because young people usually do not recognize thirst and they often haven't got an easy access to water 3.

Scientific evidence proves that a soft dehydration, as a loss 1 % of body weight, can cause reduction of concentration and cognitive performance with consequences on memory and attention in children.4,5

An English systematic study about school policies on drinking water 4 compared three different contexts: schools in which water in the classroom was prohibited, schools that allowed limited access to water (for example, the water was allowed in the classroom, but not on the desk) and schools that had open access to water (for example, water was allowed in the classroom and bottles were kept at the desk). The results showed that the percentage of children who consumed less than the recommended daily amount of fluid was significantly higher in the schools that prohibited water consumption (81%) and in the schools that had limited access to water during the school day (80%). This percentage was considerably reduced in the schools where children had free access to water (46.5%). In Italian schools generally access to water is limited and water consumption is allowed only at lunch 7.

METHODS Study Design and participants

In this cluster randomized controlled pilot study, organized and managed by IRCCS Policlinico San Donato researchers, students (both male and female) aged from 12 to 14 will be enrolled.

Consent to participate in study was obtained from representatives of the school during a meeting organized before the study. All students and their parents gave informed consent to participation. The study protocol was approved by the local Ethics Committee (protocol number 159/INT/2017).

This 5-months project involves 214 middle school students (ten classes in total).

The recruited students will be randomized in two groups; both intervention and control group include five classes.

Intervention All pupils from the intervention and control classes will be taken anthropometric, blood pressure measurements and simple urine samples; a questionnaire related to dietary and physical activity habits and cognitive tests (to evaluate cognitive performances in terms of attention, memory and concentration) will be administered; the ten classes will receive changes in the school environment and individual reinforcement tools.

Changes in class environment: only in the intervention classes refillable water dispensers and water consumption poster will be placed; every class will receive 5 bottles (18 Liters/each) per week, for a total of 100 bottles to use from January to May.

Changes in the school environment: educational posters adapted from The Healthy Eating Plate conveying messages promoting healthy diet, water consumption, and daily exercise will be posted in school.

Reinforcement tools: three health and water consumption promoting lessons, held by expert nutritionists, will be included in the curriculum. Students will be received an easy textbook developed by our nutritionist team as a support to school lessons and as a tool for involving parents. A re-usable BPA-Free water bottles to encourage water consumption and a pedometer to encourage them to be physically active will be supplied.

Only in intervention classes, automated text messages promoting water consumption will be sent in the morning to students and their parents.

OUTCOME MEASURES Primary Outcome Measure: hydration status

Secondary Outcome Measure: correlation and the variation between hydration status and cognitive performances (attention, memory and concentration).

PROCEDURES Urine sample collection and cognitive tests administration will be performed at the beginning and at the end of one school day on January and on May). Anthropometric measurements and eating habits and lifestyle questionnaires will be performed before and after the intervention (on January and May).

Osmolality test: hydration status Hydration status will be evaluated through urinary osmolality test, which indicates the solute concentration to kilograms solvent ratio (mOsm/kg).

According to Katz et al.8 a value over 800 mOsm / kg indicates dehydration status, while a value lower than 800 mOsm / kg indicates normal hydration status.

Urinary osmolality test:

* It is easy to use (it is sufficient a urine sample to carry out the analysis)
* It is accurate (in terms of sensibility and specificity) and it is a valid hydration index9.

The samples will be transported at the Clinical Pathology Medicine Laboratory-1 (SMEL-1), I.R.C.C.S. Policlinico San Donato University Hospital, where they will be stored at 2-8° C until they will be analysed.

Cognitive areas evaluation protocol To evaluate the hydration status effects on cognitive performances several neuropsychological tests from the Neuropsychological Assessment Battery for Adolescence (BVN 12-18) 10 will be administrated to all students. These allow cognitive performances measurement on various domains like memory, attention, executive and visuo-spatial functions.

Tests will be administrated by clinical psychologists during an estimated time of about 60 minutes (including explanations).

Tests from BVN are composed by:

1. Involved areas: selective and sustained attention. Selective visual attention test Structure: subjects must search and indicate the same squares as the target. Available time: 3 minutes. Scoring: sum of correct answers.
2. Involved areas: Attention, logic reasoning, executive functions, calculation domain.

Reasoning test and arithmetical judgments Structure: first part of mental calculation and second part of numbering. Available time: 10 minutes. Scoring: sum of correct answers of two parts

* Involved areas: short term verbal memory, working memory Direct and reverse Digit Span Structure: test is composed of increasing series of numbers; subject must remember the series Available time: 10 minutes. Scoring: score given by the longest series for both direct span and reverse span.
* Involved areas: language; executive function. Phonetic fluency Structure: the subject must write on paper the greatest number of words starting with three different letters Available time: 1 minute for each letter for a total of 3 minutes. Scoring: sum of written words.
* Involved areas: visual perceptive functions. Street test Structure: presentation of degraded figures; subject must found the original figure and writing it on paper.

Available time: 30 second for every image for a total of 7 minutes. Scoring: sum of correct answers given within 30 seconds.

Data elaboration and statistical analysis:

Covariance analysis will be used to evaluate the variations of hydration status, comparing intervention group versus control group.

Standard error will be calculated trough a strong estimator which considers the study cluster design.

A sample size of five-classes, with about 25 students for each class, has been estimated to evaluate a difference of 0.5 standard deviation of differences in urinary osmolality in both groups (intervention and control) between morning and afternoon time; it is considered an intra-classes correlation coefficient of 0.02 and a power of 80%.

The standard deviation difference of 0.5 has been evaluated considering Fadda et al. 2012 published on Appetite.

The assessment of the sample size has been done with "cluster randomized power analysis" procedure of PASS 11.

Publication Policy:

During this pilot study, researchers are the only owners of all collected data and they will publish data in an unconditional and integral way.

ELIGIBILITY:
Inclusion Criteria:

All secondary school students aged 12-14

Exclusion Criteria:

None

Ages: 12 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 214 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-01-19 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Hydration status | Five months. From January to May.
  The hydration status is measured through urinary osmolality test, which indicates the solute concentration to kilograms solvent ratio (mOsm/kg): a value over 800 mOsm / kg indicates dehydration status, a value lower than 800 mOsm / kg indicates normal hydration status.

SECONDARY OUTCOMES:
Cognitive performance | Five months. From January to May.
  Correlation and the variation between hydration status and cognitive performances (attention, memory and concentration).

CONTACTS AND LOCATIONS:
Overall Officials: Alexis E Malavazos, MD, PhD, Principal Investigator — IRCCS Policlinico S. Donato
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Milan, Italy

IPD SHARING:
Plan to Share IPD: No